CLINICAL TRIAL: NCT04897594
Title: A Multi-Center, Randomized, Double-Blind, Dose-Ranging, Placebo-Controlled, Proof of Concept, Adaptive, Phase 1b Clinical Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of Orally Administered TERN-201 in Patients With Presumed Non-Cirrhotic Non-Alcoholic Steatohepatitis (NASH)
Brief Title: AVIATION Study: A Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy Study of TERN-201 in Patients With Non-Cirrhotic Non-Alcoholic Steatohepatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Terns, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: TERN201-1007
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2023-12

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: Vascular adhesion protein-1(VAP-1)/ semicarbazide-sensitive amine oxidase (SSAO); Nonalcoholic steatohepatitis (NASH); Nonalcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TERN-201 10mg (Experimental): Orally administered
  Interventions: Drug: TERN-201
- TERN-201 20mg (Experimental): Orally Administered
  Interventions: Drug: TERN-201
- Placebo (Placebo Comparator): Orally administered
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TERN-201 — Investigational drug
  Arms: TERN-201 10mg; TERN-201 20mg
Other: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1b multi-center, randomized, double-blind, dose-ranging, placebo-controlled, adaptive study to evaluate the safety, pharmacokinetics (PK), pharmacodynamics (PD) of TERN-201 in patients with non-cirrhotic NASH.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 75 years of age
* Overweight or obese with a body mass index (BMI) ≥ 25 kg/m2
* Presumed NASH based on clinical characteristics or prior liver biopsy
* ALT ≥ 43 IU/L for men and ≥ 28 IU/L for women
* MRI-cT1 value> 800 ms
* Written informed consent

Exclusion Criteria:

* History or clinical evidence of chronic liver diseases other than NAFLD
* History or clinical evidence of cirrhosis, hepatic decompensation or other severe liver impairment
* History of liver transplant, or current placement on a liver transplant list
* Weight loss of > 5% total body weight within 3 months prior to Screening

Note: Other protocol-defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: clinicaltrials@ternspharma.com, Study Director — Terns, Inc.
Locations (11):
- United States (11):
  - Terns Clinical Study Site 1018, Tucson, Arizona
  - Terns Clinical Study Site 1024, Tucson, Arizona
  - Terns Clinical Study Site 1004, Coronado, California
  - Terns Clinical Study Site 1039, Los Angeles, California
  - Terns Clinical Study Site 1001, Panorama City, California
  - Terns Clinical Study Site 1040, Rialto, California
  - Terns Clinical Study Site 1013, San Diego, California
  - Terns Clinical Study Site 1010, Bastrop, Louisiana
  - Terns Clinical Study Site 1006, San Antonio, Texas
  - Terns Clinical Study Site 1003, San Antonio, Texas
  - Terns Clinical Study Site 1019, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients who orally administered the Placebo
- TERN-201 10mg: Patients who orally administered 10mg of TERN-201
- TERN-201 20mg: Patients who orally administered 20mg of TERN-201
Period: Overall Study
Arm/Group | Placebo | TERN-201 10mg | TERN-201 20mg
Started | 17 | 20 | 15
Completed | 16 | 19 | 12
Not Completed | 1 | 1 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Sponsor Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TERN-201 10mg | TERN-201 20mg | Total
Number analyzed (Participants) | 17 | 20 | 15 | 52
Age, Continuous [Median (Full Range); unit: years] | 59 [27 to 68] | 49 [28 to 68] | 48 [41 to 72] | 50.5 [27 to 72]
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 13 | 18 | 13 | 44
  >= 65 years | 4 | 2 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 9 | 35
  Male | 4 | 7 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 14 | 9 | 34
  Not Hispanic or Latino | 6 | 5 | 5 | 16
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1 | 0 | 1 | 2
  Asian | 0 | 0 | 2 | 2
  Black or African American | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 15 | 18 | 10 | 43
  Other | 0 | 0 | 1 | 1
  Not Reported | 0 | 0 | 1 | 1
  Unknown | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient Incidence of Adverse Events for TERN-201 Versus Placebo
Description: Number of patients experiencing at least 1 TEAE (Safety Analysis Set). TEAE = Treatment-emergent adverse event. Please see additional details in Adverse Events section.
Time Frame: Day 1 through Week 16
Population: Safety Analysis Set consists of all patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TERN-201 10mg | TERN-201 20mg
Number analyzed (Participants) | 17 | 20 | 15
Participants | 9 | 11 | 8

2. Primary Outcome: Treatment-Emergent Laboratory Abnormalities
Description: Number of patients with any worsening of ≥ 2 NCI CTCAE Grades in each laboratory assessment category.
  CTCAE = Common Terminology Criteria for Adverse Events; NCI = National Cancer Institute; laboratory abnormalities were classified according to NCI CTCAE, version 5, Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-Threatening
Time Frame: Day 1 through Week 16
Population: Safety Analysis Set consists of all patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TERN-201 10mg | TERN-201 20mg
Number analyzed (Participants) | 17 | 20 | 15
Participants
  Serum Chemistry | 0 | 1 | 1
  Fasting Lipids | 0 | 0 | 0
  Hematology | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Day 1 through Week 16
Arm/Group | Placebo | TERN-201 10mg | TERN-201 20mg
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/20 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20 | 0/15
Other Adverse Events (participants affected / at risk) | 9/17 | 11/20 | 8/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | TERN-201 10mg (N=20) | TERN-201 20mg (N=15)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0
Steatorrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT04897594/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT04897594/SAP_001.pdf